CLINICAL TRIAL: NCT00593060
Title: A Phase I Trial of Temsirolimus (CCI-779, Torisel) Combined With Cetuximab (Erbitux) in Cetuximab-Refractory Colorectal Cancer
Brief Title: Temsirolimus (CCI-770, Torisel) Combined With Cetuximab in Cetuximab-Refractory Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeffrey W. Clark, MD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor-Investigator, Jeffrey W. Clark, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-172
Record Dates: First submitted 2007-12-28; First posted 2008-01-14 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Colorectal Adenocarcinoma
Keywords: Temsirolimus; cetuximab; metastatic disease
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — temsirolimus; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temsirolimus Combined With Cetuximab (Experimental)
  Interventions: Drug: Temsirolimus; Drug: Cetuximab

INTERVENTIONS:
Drug: Temsirolimus — Given intravenously every week of each 28-day cycle (days 1, 7, 15, 22). Participants can continue to receive study treatment as long at their tumor is responding.
  Other Names: Torisel; CCI-779
Drug: Cetuximab — One dose is given intravenously 7 days prior to the start of each 28-day cycle, then it is given every week (along with temsirolimus)of each 28-day cycle (on days 1, 7, 15, 22). Participants can continue to receive study treatment as long at their tumor is responding.
  Other Names: Erbitux

SUMMARY:
In this study, the investigational drug, temsirolimus, will be combined with cetuximab, a biologic agent used in the treatment of colorectal cancer. Cetuximab in combination with temsirolimus may be more effective in treating advanced colorectal cancer than cetuximab alone. The purpose of this research study is to try to define the highest dose of cetuximab that can be used safely in combination with temsirolimus to treat advanced colorectal cancer that has progressed through standard therapy.

DETAILED DESCRIPTION:
* Because this is a study to determine the highest dose of cetuximab that can be safely given with temsirolimus, groups of 3 participants will be treated at gradually increasing doses of cetuximab. Each group of 3 participants must complete 4 weeks (1 cycle) of treatment before the following group of 3 participants can start treatment at the higher dose.
* Cetuximab is administered intravenously 7 days before the treatment cycle begins. Participants will receive a cetuximab infusion every week of the treatment cycle (days 1, 8, 15, 22) along with temsirolimus. Temsirolimus is also given intravenously.
* As a precaution, participants will be pre-medicated with Benadryl/diphenhydramine to help prevent an allergic reaction.
* During the study participants will have weekly clinical visits. Each clinic visit will last approximately 2-3 hours. During the clinic visit, the following tests and procedures will be performed: Physical exam; vital signs; and blood tests. A CT scan will be performed after every 2 cycles (8 weeks).
* Pharmacokinetic (PK) blood samples will be taken at various points during the study. For each PK sample, we will take about 1 teaspoon of blood. There will be a total of 22 tubes of blood taken for the PK study.

ELIGIBILITY:
Inclusion Criteria:

* Previously treated metastatic colorectal adenocarcinoma, histologically proven. Subjects must have previously received and had evidence of progression on cetuximab, bevacizumab, 5FU, irinotecan, and oxaliplatin, or demonstrated intolerance to those agents (except cetuximab).
* Measurable disease by RECIST criteria
* ECOG Performance Status 0 or 1.
* Male or female, 18 years of age or older.
* Life expectancy greater than or equal to 12 weeks.
* At least 2 weeks have elapsed between previous anti-cancer therapy AND resolution of any skin rash related to prior treatment with an epidermal growth factor receptor inhibitor.
* Lab values within ranges as outlined in protocol

Exclusion Criteria:

* Diagnosis of second malignancy within the last 3 years, except for adequately treated basal cell carcinoma or squamous cell skin cancer.
* Ongoing cardiac dysrhythmias of NCI CTCAE grade >/=2, atrial fibrillation, QTc prolongation to >450msec for males and >470 msec for females.
* Known immunodeficiency disorders or active infections requiring treatment
* Pregnancy or breastfeeding
* Brain metastases, spinal cord compression, carcinomatous meningitis, or leptomeningeal disease
* Prior radiation therapy or major surgery within 2 weeks of study entry
* Prior radiation therapy to > 25% of the bone marrow
* Treatment with other experimental or alternative therapies during the course of the trial
* History of hypersensitivity to polysorbate or cetuximab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2007-11-01 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
To determine the dose-limiting toxicities and maximal tolerated doses of cetuximab combined with temsirolimus. | 2 years
To determine the dosing regimen appropriate for Phase 2 studies of the combination. | 2 years
To determine the pharmacokinetics of combined treatment with cetuximab and temsirolimus. | 2 years

SECONDARY OUTCOMES:
To document objective response rate and progression-free survival in patients treated with the combination. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey W Clark, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts